CLINICAL TRIAL: NCT01720030
Title: Prospective, Randomized, Monocenter, Double Blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Levosimendan in Intensive Care Patients With Acute Kidney Injury
Brief Title: Levosimendan in Acute Kidney Injury Study
Acronym: LAKIS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VieCuri Medical Centre (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Dr. Jos le Noble, PhD, MD, VieCuri Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Levosimendan in AKI Study
Record Dates: First submitted 2012-10-03; First posted 2012-11-01 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Acute Kidney Injury
Keywords: Renal; Acute Kidney Injury; AKI; Levosimendan; Simdax; Renal perfusion; Mortality; Renal flow
MeSH Terms: conditions — Acute Kidney Injury | interventions — Simendan; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional therapy (Placebo Comparator): Standard of care as protocolized locally
  Interventions: Drug: Conventional therapy
- Levosimendan (Experimental): The experimental group receives standard treatment supplemented by levosimendan (0.2 µg/kg/min) for 24 hours within 36 hrs following onset of AKI.
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — Verum therapy
  Other Names: Simdax (R)
  Arms: Levosimendan
Drug: Conventional therapy — Placebo therapy to safeguard blinding
  Other Names: Standard care plus placebo comparator
  Arms: Conventional therapy

SUMMARY:
We hypothesise that levosimendan will have a positive influence on renal function during acute kidney injury in adult intensive care patients.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate whether the use of levosimendan is able to improve renal function.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed adult patients with AKI

Exclusion Criteria:

* Failure to obtain written consent to participate from patient or legal representative (by deferred consent)
* Patients entering the ICU for post-operative observation with an estimated length of stay less than 24 hrs.
* Moribund patients
* Patients under the age of 18
* Pregnancy
* Patients suffering from pre-existing renal failure (elevated NGAL values without apparent rise in creatinine values)
* Renal replacement therapy initiated before admission due to Chronic Kidney Disease
* Hypersensitivity to levosimendan experienced by previous treatments
* Severe hypotension and tachycardia
* Significant mechanical obstruction affecting ventricular filling or outflow or both.
* Severe hepatic impairment (ALAT/ASAT>400U/L)
* Patients will be excluded if the treating physician judges that study participation is undesirable for medical, medical-ethical or other reasons
* Known history of Torsades de Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in renal function | Baseline and every 24 hours until end ICU stay
  Daily analysis of kidney function expressed in endogenous creatinine clearance

CONTACTS AND LOCATIONS:
Overall Officials: Jos Le Noble, MD PhD, Principal Investigator — VieCuri Medical Centre
Locations (1):
- VieCuri Medical Center, Venlo, Limburg, Netherlands